CLINICAL TRIAL: NCT04442919
Title: Influence of METHoxyflurane on ANtiplatelet Effect of Ticagrelor in Patients With Unstable Angina Pectoris - METHANE Study
Brief Title: Influence of METHoxyflurane on ANtiplatelet Effect of Ticagrelor in Patients With Unstable Angina Pectoris
Acronym: METHANE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Professor, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METHANE
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Unstable Angina
MeSH Terms: conditions — Angina, Unstable | interventions — Methoxyflurane; Ticagrelor; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ticagrelor followed with methoxyflurane (Experimental): patients who received ticagrelor followed with inhaled methoxyflurane due to unstable angina
  Interventions: Drug: Ticagrelor followed with Methoxyflurane
- Ticagrelor followed with morphine (Active Comparator): patients who received ticagrelor followed with intravenous morphine due to unstable angina
  Interventions: Drug: Ticagrelor followed with Morphine
- Ticagrelor (Active Comparator): patients who received ticagrelor without any analgesia due to unstable angina
  Interventions: Drug: Ticagrelor alone

INTERVENTIONS:
Drug: Ticagrelor followed with Methoxyflurane — patients who received ticagrelor followed with inhaled methoxyflurane due to unstable angina
  Other Names: Brilique + Penthrox
  Arms: Ticagrelor followed with methoxyflurane
Drug: Ticagrelor followed with Morphine — patients who received ticagrelor followed with intravenous morphine due to unstable angina
  Other Names: Brilique + Morphine
  Arms: Ticagrelor followed with morphine
Drug: Ticagrelor alone — patients who received ticagrelor without any analgesia due to unstable angina
  Other Names: Brilique
  Arms: Ticagrelor

SUMMARY:
The purpose of this study is to evaluate differences in the pharmacokinetics and pharmacodynamics of ticagrelor and its active metabolite in patients who received ticagrelor followed with methoxyflurane versus ticagrelor followed with morphine or ticagrelor alone due to unstable angina pectoris

DETAILED DESCRIPTION:
Results of the IMPRESSION trial published in 2015 proved that morphine use in patients with acute coronary syndromes (ACS) is associated with undesirable impact on pharmacokinetics (PK) and pharmacodynamics (PD) of ticagrelor. Despite that, morphine is still a standard analgesic treatment in ACS patients and it should not be routinely withdrawn. Based on contemporary knowledge, morphine, acting via mi-opioid receptors, was found to inhibit gastrointestinal motility or induce adverse effects such as nausea or vomiting.

We decided to design a clinical study aiming to evaluate the impact of methoxyflurane on PD of ticagrelor in patients diagnosed with unstable angina pectoris (UA). Methoxyflurane is an inhaled anesthetic, registered in Poland in emergency medicine for pain alleviation in trauma patients. The drug was widely used in 1960s to induce general anesthesia, however its clinical utility was reduced with the development of novel anesthetic agents. Taking into account its different mechanism of action, it can be presumed that, contrary to morphine, no respiratory depression should be observed as well as no attenuation or delay of antiaggregatory effect of ticagrelor should occur, as no interaction with mi-receptor in gastrointestinal tract is related to activity of methoxyflurane.

Patients will be randomized in a 1:1:1 ratio into the study arms as follows: 1) 180 mg ticagrelor (2 integral tablets of 90 mg ticagrelor) followed by 3 mg inhaled methoxyflurane, 2) 180 mg ticagrelor followed by 5 mg intravenous morphine, 3) 180 mg ticagrelor alone

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of unstable angina
* Male or non-pregnant female, aged 18-80 years
* Provision of informed consent for angiography and PCI
* GRACE score <140 pts

Exclusion Criteria:

* Treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* Current treatment with morphine or any opioid "mi" receptor agonist
* Hypersensitivity to ticagrelor
* Current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* Active bleeding
* History of intracranial hemorrhage
* Recent gastrointestinal bleeding (within 30 days)
* History of coagulation disorders
* Platelet count less than <100 x10^3/mcl
* Hemoglobin concentration less than 10.0 g/dl
* History of moderate or severe hepatic impairment
* History of major surgery or severe trauma (within 3 months)
* Risk of bradycardic events as judged by the investigator
* Second- or third-degree atrioventricular block during screening for eligibility
* History of asthma or severe chronic obstructive pulmonary disease
* Kidney disease requiring dialysis
* Manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* Respiratory failure
* History of severe chronic heart failure (NYHA class III or IV)
* Concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* Body weight below 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Mean platelet reactivity between the study arms | 6 hours
  Mean platelet reactivity between the study arms, assessed using the Multiplate Analyzer

SECONDARY OUTCOMES:
The percentage of high platelet reactivity patients (HPR) throughout the study period | 6 hours
  the percentage of patients with high platelet reactivity throughout the study period
Mean time to achieve platelet reactivity below the threshold for HPR | 6 hours
  Mean time required for patients to receive low platelet reactivity in each study arm
area under the plasma concentration-time curve for ticagrelor and its active metabolite between the study arms | 6 hours
  area under the plasma concentration-time curve for ticagrelor and its active metabolite between the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Professor, Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No